CLINICAL TRIAL: NCT05003050
Title: Energy Therapy and Meditation Based Practice to Alleviate Sleep Difficulties in Adolescents and Young Persons With Liver Disease and Liver Transplantation
Brief Title: Energy Therapy and Meditation Based Practice for Sleep Difficulties
Acronym: ET&MforSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Anju Bhatia, Principal Investigator Dr Anju Bhatia, King's College Hospital NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KingCHLDH
Record Dates: First submitted 2021-07-29; First posted 2021-08-12 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Liver Diseases
MeSH Terms: conditions — Liver Diseases | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: 3 groups each group 10 participants 10 Standard of Care Group 10 Meditation Based Practice 10 Energy Therapy (Pranic Healing)
Who Masked: Participant, Investigator
Masking Description: Randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meditation Based Group (Experimental): 8 sessions weekly for 8 weeks Each session for 1hour Sessions on line (virtual) Self-care tools and techniques, mindfulness and meditation
  Interventions: Other: Meditation
- Energy Therapy (Pranic Healing) (Experimental): 8 Sessions Weekly sessions for 8 weeks Each session 1 hour Pranic Healing (Energy Therapy)
  Interventions: Other: Pranic Healing
- Stanrd of Care Group (No Intervention): Routine medical care and appointments

INTERVENTIONS:
Other: Meditation — Holistic natural therapy
  Arms: Meditation Based Group
Other: Pranic Healing — Energy therapy
  Arms: Energy Therapy (Pranic Healing)

SUMMARY:
Sleep difficulties have been identified as one of the most distressing symptoms for adolescents with Chronic Liver Disease (CLD), Autoimmune Liver Disease (AILD) and Liver Transplantation (LT), sleep difficulties have a direct negative impact on quality of life. The underlying pathophysiological mechanisms for this are complex. In addition Adolescents with chronic illness tend to have a higher rate of mental health problems than the general population. The complexity of sleep deprivation, fatigue, stress and anxiety, may well all be contributory factors to these patients having poor adherence to their medication. This in turn has a negative impact on the success of their tissue graft or indeed increases the likelihood for transplant surgery.

Due to the risks of medication toxicity and dependency, there is a need for further research to address the issues of insomnia, stress and anxiety with a non - pharmacological approach for these Adolescent chronically ill patients. Meditation Based Practices and Energy Therapies (Acupuncture) have gained robust scientific evidence over the last 20 years to demonstrate their efficacy for patients with insomnia, stress and anxiety.

This study aims to demonstrate the benefits of a non - touch Energy Therapy (ET) and a Meditation Based Practice (MBP) to relieve symptoms of insomnia, stress and anxiety in Adolescents with CLD, ALD and LT. The participants will be 16 - 24 years old. The intervention will have 3 groups, Standard of Care Group, MBP and ET. The intervention will be for 8 weeks with the ET and MBP group each receiving 1 hour of therapy each week for 8 weeks. The data will be collected with questionnaires and actigraph wrist devices.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE The liver is a vital organ responsible for enabling our body to digest food and rid itself of toxic substances. There are more than 100 types of liver disease affecting both children and adults presenting with a wide variety of symptoms. Young people (YP) with chronic illness tend to have a higher rate of mental health problems compared to the general population, with psychosocial complex issues affecting adherence to medication and resulting poorer health outcomes. Adolescents that have liver transplants (LT) demonstrate an inferior success rate compared to children and adults across all solid organ transplant groups.

This seems to be partially attributed to the high rate of non - adherence to medication which is a common issue amongst this age group.

Adolescence is the peak time for the onset of mental health problems with approximately 50% of mental health illnesses appearing before the age of 14 years and 75% of mental health problems developing before the age of 24 years.

Rates of anxiety, depression and behaviour difficulties are further elevated in children and adolescents with physical health problems.

A diagnosis of Autoimmune liver disease (ALD) between the ages of 14 - 20 years has been found to be independently predictive of liver related death or the need for liver transplantation compared with other age groups. In view of organ shortages, avoiding transplantation in these patients is a priority and focus on non - adherence (NA) to medication in patients with ALD. The focus on minimising NA in ALD aims to prevent avoidable transplantation and after LT aims to reduce graft loss.

Hames aimed to identify from a large cohort of YP who had already received a LT having had ALD and CLD their prevalence rates of anxiety and depression and factors associated with this.

These patient's demonstrated, psychological stresses worry (30.2 %) and low self - esteem (27.5%) among physical complaints almost 50% cited fatigue. Nearly 33% of participants also cited sleep difficulties.

Sleep difficulties have been identified as one of the most distressing symptoms for adolescents with LT and they are negatively correlated with health related quality of life in both children and adolescents. It has been, suggested psychological interventions for sleep problems are highly effective and should be evaluated for this population as a priority. Patients with CLD or patients who have had LT both cohorts exhibit sleep difficulties.

Due to the potential for medication toxicity in these disabled patients further studies are needed to address the potential role of non - drug therapies (eg. CBT, mindfulness, yoga). It is not, recommended for these young people with chronic illness to then take medication for insomnia due to toxicity risks.

Insomnia and fatigue will affect school, home life, medical health and medication adherence. There therefore is a true clinical need for complementary therapies to be considered.

Meditation and Energy associated therapies have shown efficacy with patients that have chronic illness/ pain /insomnia. These complimentary therapies are often Eastern in origin however during the last 30 years these therapies have been practiced and researched widely in the UK, demonstrating efficacy in multiple dimensions.

Meditation and Energy Therapy Meditation can be defined as a family of complex emotional and attentional regulatory training regimes - developed for various ends including the cultivation of wellbeing and emotional balance.

There has been an explosion of interest in mindfulness based programs such as Mindfulness based stress reduction program (MBSR) and mindfulness based cognitive therapy (MBCT) in the last 2 decades.

MBSR has accrued a robust evidence base in improving mental health outcomes in those with chronic physical health problems. MBCT is an adaptation of the MBSR program, developed to teach those at risk of depressive relapse, skills to stay well and has been shown to be effective.

The durability of the MBSR program is notable, benefits have been obtained with no evidence of adverse events with these findings, suggesting clinicians should consider recommending MBSR to transplant recipients that are affected by these symptoms particularly anxiety and poor sleep.

Those with chronic illness such as ALD and LT are more susceptible to stress and anxiety and a higher prevalence of S&A and depression in YP and is demonstrated by Hames at King's College Hospital London. .

Although in its infancy in the 'Western World, Energy therapies are demonstrating they can help as a valuable adjunct to traditional medical practices to enhance the recovery process of patients.

Of the family of energy therapies Acupuncture is the first wave, acupuncture is widely practiced globally and within the UK and the NHS, for 30 years.

Similar to acupuncture Pranic Healing is an Energy Therapy with fundamental, principles and beliefs akin to those in acupuncture.

This Energy Therapy is based on the principle that energy flows freely throughout the body via channels and again similarly to acupuncture, energy is removed from specific points around the affected area that has stagnated energy and often causing pain. Removal of this energy enables free flow to again resume and recovery to occur. Pranic Healing similar to acupuncture follows exact protocols for each condition. It is a non - touch systematic therapy. For each physiological and psychological condition there is an exact protocol that must followed precisely for the treatment to be effective.

Acupuncture has proved itself to be effective for many chronic illnesses as an adjunct to traditional medical practice and has been recognised as an alternative medical therapy for insomnia.

As there is a real need to provide complementary non pharmacological therapy for YP with liver disease, insomnia and its associated difficulties. T'his study is justified in evaluating 2 complementary therapies that are non-pharmacological, akin in approach to recognised and utilised complementary therapies already in practice in the NHS (MBSR and Acupuncture ) The aspiration being that YP with ALD / LT suffering with insomnia, stress and anxiety will have improvements in their symptoms in turn improving their quality of life and adherence to medication.

OBJECTIVES Primary Objective

* To give these patients an opportunity to experience a therapy that is non - pharmacological
* To experience inner peace and relaxation during these sessions
* To improve sleep quality for these patients
* To reduce stress and anxiety within the body
* To reduce fatigue

Secondary Objectives

* To improve their overall wellbeing
* To encourage them to feel more positive within their lives
* To improve their adherence to medication

STUDY DESIGN DESIGN AND METHODOLOGY This study is an experimental, longitudinal study designed to evaluate the efficacy of 2 non pharmacological complementary therapies for patients with ALD, CLD, LT, sleep difficulties, stress and anxiety.

PARTICIPANT SAMPLE All participants are registered patients at King's College Hospital Paediatric liver, GI and Nutrition Centre.

Sample size 10 patients for each group - 3 groups Both genders Ages 16- 24 years All participants will have received a LT or have some form of CLD and will be selected from the KCH patient data base, all interviews and treatment sessions will be conducted at KCH.

Patients will receive an information letter and patient participation sheet via post. Interested participants will have a one - hour information session.

Patients that are eligible will then have baseline characteristics assessed and be allocated to one of the 3 participant groups.

Meditation Based Practice Energy Therapy -Pranic Healing Standard of Care

All participants will continue with their routine care, medication and treatment at KCH. The, three groups will run parallel and independent of each other.

This is a randomised control trial. BASELINE CHARACTERISTICS -will be, taken prior to the intervention. PARTICIPANT INFORMATION - participation information sheet, an information booklet explaining what will happen during the intervention, a sleep hygiene information sheet, Actigraphy watches (Fitbit). Participants will be requested to wear this for 2 weeks prior to the intervention, throughout the intervention and for 2 weeks afterwards and again at 3 months for 2 weeks.

DATA COLLECTION Subjective data - Questionnaires, sleep diary and calendar for both groups. Questionnaires - will be completed prior to the intervention, at the end of 8 weeks and again at 3 months The IMPARTS (Integrated mental and physical healthcare Research: Training Services) System contains a core set of measures, these will form part of the questionnaires in this study.

1. PHQ9
2. GAD7
3. BIPQ
4. PSQI Assesses 7 domains of sleep - quality, latency, duration, efficiency, disturbances, benefit of sleep medication and daytime dysfunction Sleep diary - A sleep diary is attached, participants to complete each morning for 8 weeks Objective data Actigraphy - To record sleep, and record movements that can be used to estimate sleep parameters. Measurements will be TST - total sleep time WASO- wake after sleep onset. Deep sleep and light Sleep.

MEDICATION - Documentation of patient's medication dose and frequency prior to intervention will be recorded and continue in the normal way.

RANDOMISATION - Participants will be, randomly allocated to one of the three groups.

30 blank envelopes, within each will have one of the three groups stated

* Meditation Based practice - Pranic Healing - Standard of Care The envelopes will be sealed and blank. Placed into a closed box. Recruitment lead will pick out an envelope for the participants and they will be, allocated to the group named on the inside of the envelope. Once participants have been, allocated to one of the three groups, they will then, be given the relevant information and support.

SESSION DESIGN MEDITATION BASED PRACTICE Participants will meet the meditation teacher prior to the intervention and have the opportunity to ask any questions. They will be given booklets explaining the techniques and benefits of the techniques which the will be carried out in each session.

Home practice in between sessions is encouraged, with CDs of the meditations. Each session will be one hour each week, the sessions will be online/virtual for 8 consecutive weeks.

Participants will be, given sleep diaries to complete each morning and actigraph watches The sessions will always contain the same elements. There will be 3- 5 participants in each group PRANIC HEALING Participants will have the opportunity to meet the therapist prior to the intervention and have the opportunity to ask any questions.

Participants will be, given a booklet explaining energy therapy and its benefits, a calendar with the dates and times of the sessions, sleep diaries to complete each morning, actigraph watches.

The session will be one hour each week for 8 weeks consecutively The session will be 1:1 Participant will sit in a comfortable chair The therapist will carry out exact protocols for sleep, stress and anxiety. The treatment session is painless, non - invasive and non- touch. STANDARD OF CARE Participants will have their data recorded in the same way as above. Routine medical care will continue with no intervention. All will be offered both therapies after 8 weeks of study.

ELIGIBILITY:
Inclusion Criteria:

- 16- 24 years old

Liver Disease/ Liver transplantation

Sleep Difficulties

Exclusion Criteria:

Unable to follow instruction

Severe psychological illness

Current or recent participation in a research study

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Total sleep time | 22 weeks
  Actigraph measures - Total sleep time (Mins)
wake after sleep onset | 22 weeks
  Actigraph - Wake after sleep time (mins)
deep and light sleep | 22 weeks
  Actigraph - deep and light sleep (mins)
Insomnia | 22 weeeks
  Qualitative questionnaire - Pittsburgh Sleep Quality Index (PSQI) minimum score 0 maximum score 27 higher score indicates worse sleep quality

SECONDARY OUTCOMES:
stress and anxiety | 22 weeks
  Generalised Anxiety Disorder Assessment (GAD-7) validated questionnaire Minimum score 0 Maximum score 21 higher score indicates high levels of anxiety
Perception of illness | 22 weeks
  Brief Illness Perception questionnaire (BIPQ)validated questionnaire higher score reflects a more threatening view of the illness
Depression | 22 weeks
  Patient Health Questionnaire -9 (PHQ-9) validated questionnaire minimum score 0 maximum score 27 higher score indicates increased severity of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Anil Dhawan, MD FRCPCH, Study Director — Director Research and Innovation King's College Hospital
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No